CLINICAL TRIAL: NCT01124617
Title: Phase II Study of JNS024ER in Japanese Subjects With Chronic Pain Due to Diabetic Neuropathic Pain or Postherpetic Neuralgia
Brief Title: A Phase 2 Study of Tapentadol Extended-Release (JNS024ER) ) in Japanese Participants With Chronic Pain Due to Diabetic Neuropathic Pain or Postherpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017002; JNS024ER-JPN-N22
Record Dates: First submitted 2010-04-22; First posted 2010-05-17 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Pain; Diabetic Neuropathies; Neuralgia; Postherpetic Neuralgia
Keywords: Chronic pain; Diabetic Neuropathic Pain; Neuralgia, Postherpetic; Tapentadol hydrochloride extended-release; JNS024ER; Placebo
MeSH Terms: conditions — Pain; Diabetic Neuropathies; Neuralgia; Neuralgia, Postherpetic; Chronic Pain | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol (Experimental): Tapentadol hydrochloride extended-release(ER) will be administered as oral tablet at dose ranging from 25 milligram (mg) to 250 mg twice daily for 12 weeks.
  Interventions: Drug: Tapentadol
- Placebo (Placebo Comparator): Matching Placebo will be administered as oral tablet at dose ranging from 25 mg to 250 mg twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tapentadol — Tapentadol hydrochloride extended-release(ER) will be administered as oral tablet at dose ranging from 25 milligram (mg) to 250 mg twice daily for 12 weeks.
  Other Names: JNS024ER
  Arms: Tapentadol
Drug: Placebo — Matching Placebo will be administered as oral tablet at dose ranging from 25 mg to 250 mg twice daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of tapentadol extended-release (ER) tablets in Japanese participants with moderate to severe chronic (lasting a long time) pain due to painful diabetic peripheral neuropathy (pain in the extremities related to diabetes-induced nerve damage) or postherpetic neuralgia (pain lasting after condition has healed).

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), multi-center (when more than one hospital or medical school team works on a medical research study), double-blind (neither physician nor participant knows the name of the assigned drug), placebo-control (participants are randomly assigned to a test treatment or to an identical-appearing treatment that does not contain the test drug), and parallel-group (each group of participant will be treated at the same time) comparison study in Japanese participants with chronic pain due to painful diabetic peripheral neuropathy or postherpetic neuralgia. The duration of study will be 14 weeks. The study consists of 3 parts: Screening (1 Week before study commences on Day 1); Treatment (12 weeks and will include titration period [from the initiation of the study treatment to determination of the individual's maintenance dose] and maintenance period [from completion of the titration period up to12 week]); and Follow-up (1 Week). Tapentadol hydrochloride ER oral tablet or matching placebo will be administered twice daily for 12 weeks. Efficacy of the participants will primarily be evaluated through Numerical Rating Scale (NRS). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic pain due to painful diabetic neuropathy or postherpetic neuralgia continuing for at least 12 weeks before consent
* Participants with adjuvant analgesics (antidepressants, antiepileptics and diabetic peripheral neuropathy drugs) or non-opioid treatment and dissatisfied with current treatment (in sense of efficacy and/or safety) for at least consecutive 14 days during the 12 weeks before consent
* Participants have not experienced treatment with conventional opioids, except for the following cases: Short term use of opioid analgesics for treatment of post-operative acute pain more than 30 days before consent; and temporal use of codeine phosphate or dihydrocodeine phosphate for purposes other than pain relief (for example, for antitussive) more than 2 days before consent
* Mean pain intensity score of greater than or equal to 5 on an 11-point Numerical Rating Scale during 48 hours before consent and the Investigator or Sub-investigator considers that the participant should be treated with an opioid analgesic
* HbA1c within 4 weeks before consent less than or equal to 11percent (in participants with diabetic neuropathic pain)

Exclusion Criteria:

* Participants have been treated or treated with a monoamine oxidase inhibitor within 14 days before consent
* Current or a history of epilepsy or convulsive disorders or hypersensitivity to opioid analgesics
* Suggested of intracranial hypertension (for example, traumatic encephalopathy)
* Participants who have complicated condition with uncontrolled or clinically significant arrhythmia, or neuropsychiatric disorders
* Participants with moderately to severely impaired hepatic function, or severely impaired renal function

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (31):
- Japan (31):
  - Chigasaki
  - Chūōku
  - Fukuoka
  - Inashiki
  - Isesaki
  - Izumisano
  - Kanuma
  - Katsushika-ku
  - Kawaguchi
  - kooriyama
  - Kurume
  - Kyoto
  - Matsue
  - Matsumoto
  - Minatoku
  - Mitaka
  - Nagano
  - Nagoya
  - Obihiro
  - Ohta-Ku
  - Ohtsu
  - Okayama
  - Omuta
  - Osaka
  - Sapporo
  - Sendai
  - Setagaya City
  - Shimotsuga
  - Tokyo
  - Ube
  - Yokohama

RESULTS

PARTICIPANT FLOW:
Groups:
- Tapentadol: Tapentadol hydrochloride extended-release(ER) was administered as oral tablet at dose ranging from 25 milligram (mg) to 250 mg twice daily for 12 weeks.
- Placebo: Matching Placebo was administered as oral tablet at dose ranging from 25 mg to 250 mg twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Tapentadol | Placebo
Started | 60 | 31
Completed | 41 | 25
Not Completed | 19 | 6
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 9 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol | Placebo | Total
Number analyzed (Participants) | 60 | 31 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (12.98) | 68.6 (11.60) | 65.9 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 40
  Male | 34 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Numerical Rating Scale (NRS) Score at Week 12
Description: Participants were asked to assess the average pain intensity on an 11-point NRS ranging from 0 (no pain) to 10 (maximum pain imaginable) by selecting a number on the scale applicable to their pain. Baseline pain score is defined as the average pain intensity score over the last 3 days prior to the randomization. Change from Baseline in NRS score is the mean NRS score at Week 12 minus mean NRS score at Baseline.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) included all the randomly assigned participants who received at least 1 dose of study drug and had at least 1 post-randomization efficacy data. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Baseline | 6.7 (1.15) | 6.9 (1.35)
  Change at Week 12 | -2.6 (2.23) | -2.6 (2.65)

2. Secondary Outcome: Change From Baseline in Average Numerical Rating Scale (NRS) Score at Week 1 to 11
Description: Participants were asked to assess the average pain intensity on an 11-point NRS ranging from 0 (no pain) to 10 (maximum pain imaginable) by selecting a number on the scale applicable to their pain. Baseline pain score is defined as the average pain intensity score over the last 3 days prior to the randomization. Change from Baseline in NRS score is the mean NRS score at corresponding week minus mean NRS score at Baseline.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11
Population: FAS included all the randomly assigned participants who received at least 1 dose of study drug and had at least 1 post-randomization efficacy data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Change at Week 1 | -0.7 (1.15) | -0.2 (0.52)
  Change at Week 2 | -1.1 (1.47) | -0.9 (1.47)
  Change at Week 3 | -1.5 (1.75) | -1.1 (1.59)
  Change at Week 4 | -1.8 (1.88) | -1.6 (1.78)
  Change at Week 5 | -2.1 (1.87) | -1.7 (2.09)
  Change at Week 6 | -2.3 (1.97) | -2.0 (2.41)
  Change at Week 7 | -2.3 (2.10) | -2.2 (2.55)
  Change at Week 8 | -2.4 (2.12) | -2.4 (2.50)
  Change at Week 9 | -2.5 (2.20) | -2.4 (2.56)
  Change at Week 10 | -2.6 (2.22) | -2.6 (2.51)
  Change at Week 11 | -2.6 (2.25) | -2.4 (2.66)

3. Secondary Outcome: Percentage of Participants With Treatment Response Based on Numerical Rating Scale (NRS)
Description: Percentage of participants with treatment response in mean NRS score by greater than equal to 30 or 50 percent (%) in the last week from baseline were considered as responders. Participants were asked to assess the average pain intensity on an 11-point NRS ranging from 0 (no pain) to 10 (maximum pain imaginable) by selecting a number applicable to their pain on the scale.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Percentage of participants
  Greater than or equal to 30% treatment response | 48.3 | 41.9
  Greater than or equal to 50% treatment response | 33.3 | 38.7

4. Secondary Outcome: Number of Participants With Categorical Scores on Patient's Global Impression of Change (PGIC) Scale
Description: The PGIC is a 7-point scale that requires the participants to assess how much their illness has improved or worsened relative to a Baseline state at the beginning of the intervention. The response options are 1 = very much improved, 2 = much improved, 3 = minimally improve, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Week 8 and Week 12
Population: FAS included all participants who received study drug & had at least 1 post-randomization efficacy data. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure & 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 46 | 26
Participants
  Week 8: Very Much Improved (n = 46, 26) | 7 | 4
  Week 8: Much Improved (n = 46, 26) | 16 | 7
  Week 8: Minimally Improved (n = 46, 26) | 16 | 10
  Week 8: No Change (n = 46, 26) | 6 | 2
  Week 8: Minimally Worse (n = 46, 26) | 1 | 2
  Week 8: Much Worse (n = 46, 26) | 1 | 1
  Week 8: Very Much Worse (n = 46, 26) | 0 | 0
  Week 12: Very Much Improved (n = 40, 25) | 6 | 2
  Week 12 : Much Improved (n = 40, 25) | 18 | 9
  Week 12 : Minimally Improved (n = 40, 25) | 13 | 11
  Week 12 : No Change (n = 40, 25) | 2 | 2
  Week 12 : Minimally Worse (n = 40, 25) | 0 | 0
  Week 12 : Much Worse (n = 40, 25) | 1 | 1
  Week 12 : Very Much Worse (n = 40, 25) | 0 | 0

5. Secondary Outcome: Number of Participants With Categorical Scores on Physician's Global Assessment Scale
Description: Physician's Global Assessment Scale assesses the therapeutic efficacy (effectiveness) of the study drug for pain control on a 2-point scale of "effective" and "ineffective".
Time Frame: Week 8 and Week 12
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 46 | 26
Participants
  Week 8: Effective (n = 46, 26) | 41 | 19
  Week 8: Ineffective (n = 46, 26) | 5 | 7
  Week 12: Effective (n = 40, 25) | 35 | 20
  Week 12 : Ineffective (n = 40, 25) | 5 | 5

6. Secondary Outcome: Change From Baseline in Pain Interference Subscale Score Based on Brief Pain Inventory (Short Form) (BPI-sf) Scale
Description: The BPI-sf consists of 15 Items (Item 1:presence of pain; Item 2:pain location; Items 3 to 6:pain severity; Item 7:status of pain treatment; Item 8:efficacy of pain treatment; and Items 9a to 9g: interference of pain with daily life). Pain interference sub-scale score ranges from 0 (do not interfere) to 10 (completely interferes). Higher scores indicates worsening. Total score is defined as the mean scores from Items 3, 4, 5, 6 and 9 recorded on an 11-point scale where 0 = no pain and 10 = pain as bad as you can imagine. Lower score indicates an improvement in pain.
Time Frame: Baseline and Week 12
Population: FAS included all participants who received study drug & had at least 1 post-randomization efficacy data. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Baseline (n=60, 31) | 4.7 (2.13) | 4.6 (2.20)
  Week 12 (n=25,40) | -2.6 (1.92) | -2.1 (2.48)

7. Secondary Outcome: Change From Baseline in Pain Subscale Score Based on Brief Pain Inventory (Short Form) (BPI-sf) Scale
Description: The BPI-sf consists of 15 Items (Item 1:presence of pain; Item 2:pain location; Items 3 to 6:pain severity; Item 7:status of pain treatment; Item 8:efficacy of pain treatment; and Items 9a to 9g: interference of pain with daily life). Pain Sub-scale score ranges from 0 (absent [no pain]) to 10 (extreme [pain as bad as you can image]). Higher scores indicates worsening. Total score is defined as the mean scores from Items 3, 4, 5, 6 and 9 recorded on an 11-point scale where 0 = no pain and 10 = pain as bad as you can imagine. Lower score indicates an improvement in pain.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Baseline (n=60, 31) | 6.2 (1.19) | 6.3 (1.22)
  Week 12 (n=25,40) | -3.0 (1.72) | -2.6 (2.35)

8. Secondary Outcome: Change From Baseline in Brief Pain Inventory (Short Form) (BPI-sf) Total Score at Week 12
Description: The BPI-sf consists of 15 Items (Item 1:presence of pain; Item 2:pain location; Items 3 to 6:pain severity; Item 7:status of pain treatment; Item 8:efficacy of pain treatment; and Items 9a to 9g: interference of pain with daily life). Total score is defined as the mean scores from Items 3, 4, 5, 6 and 9 recorded on an 11-point scale where 0 = no pain and 10 = pain as bad as you can imagine. Lower score indicates an improvement in pain.
Time Frame: Baseline and Week 12
Population: FAS included all the randomly assigned participants who received at least 1 dose of study drug and had at least 1 post-randomization efficacy data. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Baseline (n=60,31) | 5.2 (1.58) | 5.2 (1.52)
  Change at Week 12 (n=40,25) | -2.7 (1.64) | -2.3 (2.29)

9. Secondary Outcome: Change From Baseline in Sleep Latency Based on Sleep Questionnaire at Week 12
Description: Sleep Latency was related to "How long after bedtime or lights out did the participant fall asleep last night ". Decrease in time indicates an improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 30
Minutes
  Baseline (n=60, 30) | 45.4 (65.78) | 34.7 (28.62)
  Change at Week 12 (n=40, 24) | -11.1 (49.15) | -3.1 (30.17)

10. Secondary Outcome: Change From Baseline in Time Slept Based on Sleep Questionnaire at Week 12
Description: Time slept was related to "How long did the participant sleep last night". The mean change for the time in hours slept during the last night was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Hours
  Baseline (n=60, 31) | 5.8 (1.29) | 6.4 (1.97)
  Change at Week 12 (n=40,25) | 0.3 (1.71) | 0.3 (1.58)

11. Secondary Outcome: Number of Participants With Awakenings Based on Sleep Questionnaire
Description: Number of awakenings was related to "How many times did the participant wake up during the night". Lesser number signifies better sleep.
Time Frame: Baseline and Week 12
Population: FAS included all the randomly assigned participants who received at least 1 dose of study drug and had at least 1 post-randomization efficacy data. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 30
Participants
  Baseline: 0 awakening (n=60,30) | 17 | 3
  Baseline: 1 awakening (n=60,30) | 16 | 9
  Baseline: 2 awakenings (n=60,30) | 10 | 10
  Baseline: 3 awakenings (n=60,30) | 8 | 6
  Baseline: 4 awakenings (n=60,30) | 5 | 1
  Baseline: > or = 5 awakenings (n=60,30) | 4 | 1
  Week 12 : 0 awakening (n=40,25) | 12 | 3
  Week 12 : 1 awakening (n=40,25) | 14 | 8
  Week 12 : 2 awakenings (n=40,25) | 9 | 7
  Week 12 : 3 awakenings (n=40,25) | 1 | 4
  Week 12 : 4 awakenings (n=40,25) | 3 | 2
  Week 12 : > or = 5 awakenings (n=40,25) | 1 | 1

12. Secondary Outcome: Number of Participants With Response Based on Overall Quality of Sleep Questionnaire
Description: Participants rated the overall quality of sleep last night as excellent, good, fair and poor.
Time Frame: Baseline and Week 12
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Participants
  Baseline: Excellent (n=60,31) | 0 | 1
  Baseline: Good (n=60,31) | 35 | 12
  Baseline: Fair (n=60,31) | 22 | 16
  Baseline: Poor (n=60,31) | 3 | 2
  Week 12 : Excellent (n=60,31) | 4 | 0
  Week 12 : Good (n=40,25) | 28 | 17
  Week 12 : Fair (n=40,25) | 6 | 8
  Week 12 : Poor (n=40,25) | 2 | 0

13. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey Version 2 (SF-36v2) Scores at Week 12
Description: The SF-36v2 is 36-item form related to 8 health concepts (physical functioning, role physical, role emotional, general health, social functioning, bodily pain, vitality, mental health) and 2 summary scores (physical and mental component summary). Physical functioning, role physical and bodily pain contribute to physical component; role emotional, social functioning and mental health contribute to mental component; and social functioning, vitality, and general health contribute to both. All scores are based on a scale from 0 to 100, with higher scores defining more favorable health state.
Time Frame: Baseline and Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol | Placebo
Number analyzed (Participants) | 60 | 31
Units on a scale
  Physical Functioning: Baseline (n=60,31) | 68.6 (21.88) | 61.0 (24.20)
  Role-Physical: Baseline (n=60,31) | 70.1 (27.95) | 64.3 (28.15)
  Bodily Pain: Baseline (n=60,31) | 36.2 (16.74) | 38.8 (14.50)
  General Health: Baseline (n=60,31) | 45.7 (16.73) | 44.7 (17.51)
  Vitality: Baseline (n=60,31) | 48.8 (23.49) | 50.4 (22.47)
  Social Functioning: Baseline (n=60,31) | 72.9 (26.66) | 80.2 (27.72)
  Role-Emotional: Baseline (n=60,31) | 68.9 (30.91) | 68.5 (28.19)
  Mental Health: Baseline (n=60,31) | 57.6 (24.54) | 61.8 (22.04)
  Mental Summary: Baseline (n=60,31) | 43.9 (12.27) | 47.6 (10.65)
  Physical Summary: Baseline (n=60,31) | 36.0 (16.11) | 31.7 (16.48)
  Physical Functioning: Change at Week 12 (n=40,25) | 5.4 (13.65) | 4.8 (14.89)
  Role-Physical: Change at Week 12 (n=40,25) | 6.6 (21.74) | 4.8 (22.26)
  Bodily Pain: Change at Week 12 (n=40,25) | 10.5 (15.43) | 7.0 (15.57)
  General Health: Change at Week 12 (n=40,25) | -0.4 (10.74) | 0.2 (11.83)
  Vitality: Change at Week 12 (n=40,25) | 9.4 (19.09) | 6.8 (22.31)
  Social Functioning: Change at Week 12 (n=40,25) | 8.1 (21.47) | 2.0 (37.27)
  Role-Emotional: Change at Week 12 (n=40,25) | 6.0 (27.02) | 5.7 (25.65)
  Mental Health: Change at Week 12 (n=40,25) | 7.8 (17.02) | 9.0 (23.98)
  Mental Summary: Change at Week 12 (n=40,25) | 4.5 (7.85) | 3.3 (11.48)
  Physical Summary: Change at Week 12 (n=40,25) | 4.4 (11.22) | 2.8 (11.56)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Tapentadol | Placebo
Serious Adverse Events (participants affected / at risk) | 4/60 | 3/31
Other Adverse Events (participants affected / at risk) | 52/60 | 26/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (N=60) | Placebo (N=31)
Urinary tract infection (Infections and infestations) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (N=60) | Placebo (N=31)
Nasopharyngitis (Infections and infestations) | 7 | 4
Gastroenteritis (Infections and infestations) | 3 | 1
Cystitis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Listless (Psychiatric disorders) | 1 | 0
Somnolence (Nervous system disorders) | 17 | 3
Dizziness (Nervous system disorders) | 5 | 2
Headache (Nervous system disorders) | 4 | 2
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Radial nerve palsy (Nervous system disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 1
Chalazion (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Trichiasis (Eye disorders) | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 19 | 0
Constipation (Gastrointestinal disorders) | 16 | 0
Vomiting (Gastrointestinal disorders) | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 5 | 0
Thirst (General disorders) | 5 | 0
Malaise (General disorders) | 3 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Blood urine present (Investigations) | 3 | 0
Liver function test abnormal (Investigations) | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 1 | 1
Protein urine present (Investigations) | 2 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Eosinophil percentage increased (Investigations) | 0 | 1
Lymphocyte percentage decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other